CLINICAL TRIAL: NCT02015338
Title: Comparing the Location of the Motor Cortex in Children Using Two Methods: EEG and TMS
Brief Title: Comparing the Location of the Motor Cortex in Children Using Two Methods
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1311M45303
Record Dates: First submitted 2013-12-04; First posted 2013-12-19 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Congenital Hemiparesis
Keywords: Hemiparesis; Cerebral Palsy; Congenital Stroke; Congenital Infarct
MeSH Terms: conditions — Paresis; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Typically Developing Children: Children with typical development (e.g. no presence of neurological disorders or diagnoses)
- Children with Hemiparesis: Children diagnosed with Hemiparesis

SUMMARY:
Hypothesis: In typically developing children (TDC), use of conventional EEG landmarks to determine the brain area that controls hand function will not differ from TMS-guided determination of individual motor hotspots. In children with hemiparesis, however, those two locations will diverge. The prediction is that TMS will best guide Transcranial Direct Current Stimulation (tDCS) interventions

DETAILED DESCRIPTION:
Congenital hemiparesis, mainly due to stroke, affects approximately 25% of children with cerebral palsy. Noninvasive brain stimulation has emerged to influence improvements in hand function specifically in children with congenital hemiparesis due to stroke.

The use of one type of noninvasive brain stimulation, Transcranial Direct Current Stimulation (tDCS), in conjunction with rehabilitation training intervention for a child with hemiparesis proposes a synergistic approach to improving hand function. Application of electrodes over certain targeted areas are placed with the intent to stimulate and influence neuronal activity.

Our preliminary evidence suggests that in children with hemiparesis due to stroke, the area for placement is variable as noted by electroencephalogram (EEG) and Transcranial Magnetic Stimulation (TMS) measurement methods, influencing the site location of optimal stimulation for tDCS.

Due to this variation, the optimal site of stimulation warrants investigation for the optimal placement of tDCS.

ELIGIBILITY:
Inclusion Criteria:

Typically Developing Children:

* Ages 8-17

Children with congenital hemiparesis due to hemispheric stroke:

* Ages 8-17
* Equal of greater than 10 degrees of active motion at the metacarpophalangeal joint
* No evidence of seizure activity within the last 2 years.

Exclusion Criteria:

Typically Developing Children:

* neurologic disorders
* indwelling metal
* pregnancy
* history of seizures

Children with hemiparesis:

* Metabolic disorders
* Neoplasm
* Epilepsy
* Disorders of cellular migration and proliferation
* Expressive aphasia
* Pregnancy
* Indwelling metal
* Botulinum toxin or phenol intramuscular block within the one-month preceding TMS application.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with congenital hemiparesis and typically developing children
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determine the location of the motor cortex by two different means | 1 year
  Determine the location of the motor cortex through two means: 1) The international 10/20 EEG system of measurement and 2) Transcranial Magnetic Stimulation (TMS) testing of cortical excitability in typically developing children and children with hemiparesis.

SECONDARY OUTCOMES:
Measurement of distance in centimeters between the 10/20 EEG C3 or C4 location and the TMS-derived motor hotspot. | 1 year
  Compare the two locations (in each hemisphere) determined by 10/20 EEG system and Transcranial Magnetic Stimulation (TMS) testing and measure in centimeters differences between the two locations.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette T Gillick, PhD, MSPT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Rich TL, Menk JS, Rudser KD, Chen M, Meekins GD, Pena E, Feyma T, Bawroski K, Bush C, Gillick BT. Determining Electrode Placement for Transcranial Direct Current Stimulation: A Comparison of EEG- Versus TMS-Guided Methods. Clin EEG Neurosci. 2017 Nov;48(6):367-375. doi: 10.1177/1550059417709177. Epub 2017 May 22. PMID 28530154
- [Background] Rich TL, Menk JS, Rudser KD, Feyma T, Gillick BT. Less-Affected Hand Function in Children With Hemiparetic Unilateral Cerebral Palsy: A Comparison Study With Typically Developing Peers. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):965-976. doi: 10.1177/1545968317739997. Epub 2017 Nov 12. PMID 29130382